CLINICAL TRIAL: NCT01589263
Title: Effectiveness of OnabotulinumtoxinA (onaBoNT-A) vs Oral Tamsulosin in Men With Benign Prostatic Hyperplasia & Lower Urinary Track Symptoms (#02-10-10-05)
Brief Title: Effectiveness of onaBoNT-A vs Oral Tamsulosin in Men With BPH and LUTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIN-023-11F; 115,132 (Other: IND); H-27457 (Other: BCM IRB); NCT01567293 (obsolete NCT alias)
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Track Symptoms
Keywords: Benign Prostatic Hyperplasia; Lower Urinary Track Symptoms; BPH; LUTS
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — onabotulinum toxin A; Botulinum Toxins, Type A; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM 1: onaBoNT-A + placebo (Active Comparator): onaBoNT-A 200 U prostate injection and placebo oral capsule daily
  Interventions: Drug: onaBoNT-A + placebo; Drug: Tamsulosin + placebo
- ARM 2: Saline + Tamsulosin (Active Comparator): Placebo prostate injection (saline) and tamsulosin 0.4 mg capsule daily.
  Interventions: Drug: onaBoNT-A + placebo; Drug: Tamsulosin + placebo

INTERVENTIONS:
Drug: onaBoNT-A + placebo — 200 U prostate injection once
  Arms: ARM 1: onaBoNT-A + placebo
  Other Names: Botox
Drug: Tamsulosin + placebo — 0.4 mg capsule daily for 3 months Arms: ARM 2: Saline + Tamsulosin
  Other Names: Flomax

SUMMARY:
Benign prostatic hyperplasia (BPH) and its related symptoms are a common condition that affects nearly half of men over age 50 and 90% of men over 80. Lower urinary tract symptoms (LUTS) caused by BPH can be very troublesome, affect an individual's quality of life significantly, and are costly.

his Phase 2 clinical research trial is a double-blind, randomized, placebo-controlled, parallel-group study to compare the treatment effects of onaBoNT-A 200 U versus 0.4 mg per day of oral tamsulosin in male Veterans diagnosed with moderate to severe LUTS [American Urologic Association Symptom Score (AUASS) equal to or greater than 8] associated with BPH. A total of 74 volunteers will be recruited to participate in this clinical trial. Volunteers will include only males who are greater than 50 years of age and diagnosed with LUTS associated with BPH. They are Veterans who visit the Michael E. DeBakey Veterans Affairs Medical Center - Houston (MEDVAMC). There are no eligibility restrictions as to race or ethnicity.

DETAILED DESCRIPTION:
This proposed intervention is the first randomized clinical trial comparing the effects of onaBoNT-A prostate injection versus alpha adrenergic antagonist medication for LUTS associated with BPH. Up to this point, clinical studies using onaBoNT-A in the prostate has been limited to patient's refractory to -1 adrenoceptor blocker therapy. The study will directly compare onaBoNT-A against -1 adrenoceptor blockers as frontline therapy in a male Veteran cohort suffering from moderate to severe LUTS. Besides its obvious efficacy in patients' refractory to -1 adrenoceptor blocker therapy, onaBoNTA injection has several potential advantages over oral agents. Focal prostate injection has been shown to be safe and obviates the systemic side effects observed with -1 adrenoceptor blockers (i.e. orthostatic hypotension, sexual dysfunction). In addition, most clinical studies demonstrate a durable response to onaBoNT-A treatment exceeding 12 months. Although this study is of modest length (i.e. total 4 years), significant results could drive paradigm shifts in how LUTS associated with BPH is treated, even with regards to frontline therapy.

Although sophisticated molecular techniques (i.e. LCM with Microarray Analysis) have been used by other investigators to characterize gene profile changes with BPH and LUTS, this will be the first study examining gene profile changes in drug na ve BPH View Protocol Record patients following treatment with the -1 adrenoceptor blocker Tamsulosin or onaBoNT-A. This study is important because scant knowledge exists on the true mechanisms by which -1 adrenoceptor blockers like Tamsulosin or onaBoNT-A improve patient urinary tract symptoms and quality of life. It is clear, however, that nerves not only regulate prostate growth and function but also account for LUTS that drive patients to seek therapy. This investigation will utilize onaBoNT-A as a biological tool to identify potential novel mechanistic pathways for future investigation that will push the development of targeted therapy to benefit those patients refractory to all pharmacologic treatment. Potential inflammatory pathways or neural sensory signaling alterations induced by BPH, which are modified by onaBoNT-A or Tamsulosin to improve symptoms via gene profile changes, can be explored by expert laboratories in the Texas Medical Center. This is a highly collaborative project utilizing expertise across departments that will foster translational work from the laboratory to the patient. Although not the primary goal of this study, the investigators will also search for possible biological markers with prognostic value that could be confirmed in a future multi-center trial.

The primary objective of this Phase 2 clinical research study is to compare the efficacy of 200 U onaBoNT-A injected into the prostate versus oral tamsulosin for the treatment of lower urinary tract symptoms caused by BPH in male Veteran volunteers at the MEDVAMC. The secondary objective is to determine the impact of tamsulosin and onaBoNT-A on the pathologic parameters and RNA profiles of epithelium and stroma in BPH tissues.

Volunteers will be randomized into two groups with one receiving ona-BoNT-A injection into the prostate and an oral placebo pill taken once daily and the other group will receive a placebo injection and an oral tamsulosin pill once daily.

Volunteers will make five clinic visits and be contacted by telephone twice.

ELIGIBILITY:
Inclusion Criteria:

* Males at least 50 years of age
* American Urological Association Symptom Score greater than 8
* Voided volume greater than 125 ml
* Maximum urinary flowrate less than 15 ml/sec.
* Must agree to all procedures and willfully consented

Exclusion Criteria:

* Any prior surgical intervention or use of 5-alpha-reductase medical intervention for BPH
* Current diagnosis of acute or chronic prostatitis (which may cause LUTS that mimic BPH)
* Previous exposure to onabotulinumtoxinA
* Overactive bladder without obstructive symptoms (i.e. decrease in force of stream, hesitancy, intermittency, post-void dribbling)
* Active urinary tract disease or biopsy of the prostate within the past 6 weeks;
* Two documented urinary tract infections of any type in the past year (UTI defined as greater than 100,000 colonies per ml urine from midstream clean catch or catheterized specimen)
* Uncontrolled diabetes
* History of bladder calculi (stones)
* Penile prosthesis or artificial urinary sphincter [placement]
* Documented bacterial or acute prostatitis within the past year
* Episode of unstable angina pectoris, myocardial infarction, transient ischemic attack, or cerebrovascular accident (stroke) within the past 6 months
* Known primary neurologic conditions such as multiple sclerosis, myasthenia gravis or Parkinson's disease, or other neurological diseases known to affect bladder function
* History or current evidence of carcinoma of the prostate or bladder, pelvic radiation or surgery, urethral stricture, or bladder neck obstruction
* Cancer that is not considered cured, except basal cell or squamous cell carcinoma of the skin (cured defined as no evidence of cancer within the past 5 years)
* Any serious medical condition that is likely to impede successful completion of the study, such as certain mental disorders, hypersensitivity to onabotulinumtoxinA or anesthetics used in the study, syncope
* Daily use of a pad or device for incontinence required
* Interested in future fertility
* Postvoid Residual (PVR) greater than 350 ml
* Serum prostate specific antigen (PSA) level greater than 8 ng/ml (Hybritech). For those with a PSA between 4-8 ng/ml, the PSA elevation must be considered to be from a benign cause in the opinion of the PI. This decision can be based on PSA velocity, previous TRUS (transrectal ultrasound) biopsy, percent free PSA, or other clinical estimations in keeping with sound urologic care
* Has taken phenylephrine, pseudoephedrine, imipramine, an anticholinergic, or cholinergic medication within the past 2 weeks
* Has taken estrogen, androgen, any drug producing androgen suppression, or anabolic steroids within the past 4 months
* Taking aminoglycosides or any drug that interfere with neuromuscular transmission. Eaton-Lambert syndrome, hemophilia, hereditary clotting factors deficiency, or bleeding diathesis
* Must be off aspirin, NSAIDS, and Coumadin for 7 or more days prior to onabotulinumtoxinA injection
* Enrolled in another treatment trial for any disease within the past 30 days

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males at least 50 years of age
Enrollment: 63 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Smith, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crawford ED, Hirst K, Kusek JW, Donnell RF, Kaplan SA, McVary KT, Mynderse LA, Roehrborn CG, Smith CP, Bruskewitz R. Effects of 100 and 300 units of onabotulinum toxin A on lower urinary tract symptoms of benign prostatic hyperplasia: a phase II randomized clinical trial. J Urol. 2011 Sep;186(3):965-70. doi: 10.1016/j.juro.2011.04.062. Epub 2011 Jul 24. PMID 21791356
- [Result] Smith CP, Chancellor MB. Emerging role of botulinum toxin in the management of voiding dysfunction. J Urol. 2004 Jun;171(6 Pt 1):2128-37. doi: 10.1097/01.ju.0000127725.48479.89. PMID 15126771
- [Result] Chancellor MB, Fowler CJ, Apostolidis A, de Groat WC, Smith CP, Somogyi GT, Aoki KR. Drug Insight: biological effects of botulinum toxin A in the lower urinary tract. Nat Clin Pract Urol. 2008 Jun;5(6):319-28. doi: 10.1038/ncpuro1124. Epub 2008 May 6. PMID 18461049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 63 subjects were consented and Informed Consent was signed by all of the subjects. These subjects were selected from PI's medical clinic. PI and the CRC explained the study to these subjects but only 21 participants started the intervention.
Groups:
- ARM 1: onaBoNT-A + Placebo: onaBoNT-A 200 U prostate injection and placebo oral capsule daily
  onaBoNT-A + placebo: 200 U prostate injection once
  Arms: ARM 1: onaBoNT-A + placebo
  Tamsulosin + placebo: 0.4 mg capsule daily for 3 months Arms: ARM 2: Saline + Tamsulosin
- ARM 2: Saline + Tamsulosin: Placebo prostate injection (saline) and tamsulosin 0.4 mg capsule daily.
  onaBoNT-A + placebo: 200 U prostate injection once
  Arms: ARM 1: onaBoNT-A + placebo
  Tamsulosin + placebo: 0.4 mg capsule daily for 3 months Arms: ARM 2: Saline + Tamsulosin
Period: Overall Study
Arm/Group | ARM 1: onaBoNT-A + Placebo | ARM 2: Saline + Tamsulosin
Started | 9 | 12
Completed | 9 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM 1: onaBoNT-A + Placebo | ARM 2: Saline + Tamsulosin | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Male | 9 | 12 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
PSA [Mean (Standard Deviation); unit: ng/mL] | 1.35 (1.35) | 1.725 (1.725) | 1.5 (1.5)
Prostate Volume [Mean (Standard Deviation); unit: CC] — Normal Range : 20-30 ccs
  CC | 26.79 (26.79) | 32.33 (32.33) | 29.56 (29.56)
AUA Symptom Score [Mean (Standard Deviation); unit: units on a scale] — AUA Score Index 0 - 7 Mild 8-19 Moderate 20-35 Severe
  units on a scale | 22.92 (22.92) | 22.78 (22.78) | 22.85 (22.85)
BPH Impact Score [Mean (Standard Deviation); unit: units on a scale] — BPH Impact Score
  Minimum: 0 (No urinary condition) Maximum: 13 (Higher number indicates the urinary condition)
  units on a scale | 7.83 (7.83) | 6.11 (6.11) | 6.97 (6.97)
Bladder Function Score [Mean (Standard Deviation); unit: units on a scale] — Sum of the RDMS Questionnaire results are graded for bladder function:
  Minimum Score: 0 indicates that there is no issue with the bladder function. Maximum Score: 24 indicates the severity of the issue with the bladder function.
  units on a scale | 7.58 (7.58) | 7.44 (7.44) | 7.51 (7.51)
Erectile Function Score [Mean (Standard Deviation); unit: units on a scale] — 22-25: No erectile dysfunction, 17-21: Mild erectile dysfunction ,12-16: Mild to moderate erectile dysfunction ,8-11: Moderate erectile dysfunction, 5-7: Severe erectile dysfunction.
  units on a scale | 21.58 (21.58) | 29.56 (29.56) | 25.57 (25.57)
Ejaculation Function Score [Mean (Standard Deviation); unit: units on a scale] — On the scale of 0-35 on ejaculation score index:
  Score of 0: Is a good ejaculation score. Score of 35: Is graded as a disease severity on ejaculation score.
  units on a scale | 20.58 (20.58) | 17.44 (17.44) | 19.01 (19.01)

OUTCOME MEASURES:

1. Primary Outcome: American Urologic Association Symptom Score (AUASS)
Description: AUA Symptom Score on a scale of 0 to 35, 35 is the worse outcome and 0 is the best outcome.
Time Frame: 3 months
Population: Volunteers were randomized on a 1:1 assignment by the MEDVAMC Research Pharmacy to either: ARM 1: BoNT-A 200 U prostate injection and placebo oral capsule daily or ARM 2: Placebo prostate injection (saline) and Tamsulosin 0.4 mg capsule daily.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1: onaBoNT-A + Placebo | ARM 2: Saline + Tamsulosin
Number analyzed (Participants) | 9 | 12
score on a scale | 18.66 (0.07) | 14.16 (0.05)

ADVERSE EVENTS:
Time Frame: 19.6 month period.
Arm/Group | ARM 1: onaBoNT-A + Placebo | ARM 2: Saline + Tamsulosin
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/12
Other Adverse Events (participants affected / at risk) | 1/9 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1: onaBoNT-A + Placebo (N=9) | ARM 2: Saline + Tamsulosin (N=12)
Unrelated (Gastrointestinal disorders) | 1 (1) | 0 (0) — One patient was removed due to serious adverse event unrelated to participation in the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1: onaBoNT-A + Placebo (N=9) | ARM 2: Saline + Tamsulosin (N=12)
Unrelated (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT01589263/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT01589263/ICF_001.pdf